CLINICAL TRIAL: NCT03227874
Title: Acute Effects of Dried Apple Consumption on Metabolic Responses in Healthy Individuals
Brief Title: Effects of Dried Apple on Metabolic Responses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: San Diego State University (Other)
Responsible Party: Principal Investigator, Dr. Shirin Hooshmand, Associate professor, San Diego State University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 2040097
Record Dates: First submitted 2017-07-19; First posted 2017-07-24 (Actual); Last update posted 2017-07-24 (Actual); Status verified 2017-07

CONDITIONS: Healthy Individual

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dried apple (Experimental): diced dried apple with 55 g carbohydrate, was consumed by the participants with 220 ml of water.
  Interventions: Dietary Supplement: Dried apple; Dietary Supplement: Muffin
- Muffin (Experimental): two muffins, each with 55 g carbohydrate, was consumed by the participants with 220 ml of water.
  Interventions: Dietary Supplement: Dried apple; Dietary Supplement: Muffin

INTERVENTIONS:
Dietary Supplement: Dried apple — diced dried apple with 55 g carbohydrate, was consumed by the participants with 220 ml of water.
Dietary Supplement: Muffin — two muffins with 55 g carbohydrate, was consumed by the participants with 220 ml of water.

SUMMARY:
Metabolic syndrome is a combination of metabolic comorbidities associated with obesity, which include impaired glucose tolerance and regulation, hypertension, dyslipidemia, and increased cardiovascular disease risk. Metabolic syndrome is highly prevalent with the growing trend of obesity that characterizes the US, with 34% of adults 20 years of age and older meeting the criteria. The number of people with diabetes is expected to increase dramatically over the next decades, coinciding with rising obesity rates in many countries. Recent studies have highlighted the beneficial effects of apple and apple products in reducing the risk of chronic disease due to their rich content of fiber, nutrients and various phytochemicals. The primary objective of the proposed research is to determine the acute effect of consumption of 240 kcal servings of dried apples versus a lowfat/high fiber muffin on blood glucose, serum insulin, and fullness (satiety). The secondary objective of the proposed research is to determine the acute effect of consumption of dried apple versus a low-fat muffin on various cognitive domains. As with any organ, the brain requires nutrients to build and maintain its structure and function, in order to perform in a harmonious manner and avoid damage from aging. Epidemiological, clinical and basic research studies suggest protective effects of several classes of nutrients against cognitive decline and risk of dementia. Twenty five male and female participants between the ages of 20-45 years with a body mass index (BMI) between 18 and 25 will be recruited to participate in the study at San Diego State University. Each participant will consume both test foods, the dried apple and muffin, on two separate visits to the lab at least a week apart. The participants will come to each lab visit after a 10 hour overnight fast. After arriving at the laboratory, the participant's will complete a cognitive pre-test (Concussion Vital Signs Test Battery) consisting of eight short cognitive tests on a computer. Next After arriving at the lab, blood samples will be collected from warmed hands by finger-prick into large (250 microliter) heparinized Natelson tubes to obtain an ample blood collection for analysis of baseline plasma concentrations of glucose and insulin. The participants will then be given 5 minutes to consume the test food. Subsequent finger-prick blood samples will be collected at 15, 30, 45, 60, 90 and 120 minutes. The participants will also rate their feelings of fullness on a visual scale prior to consumption of the test food and every 15 minutes for two hours after consumption. After the completion of the finger-prick blood samples and satiety questionnaires the participants will complete a cognitive post-test which will be a different version of the cognitive pre-test battery. Concentrations of glucose will be assessed by a handheld glucose monitor as well as an enzymatic kit. Insulin will be assessed by ELISA or radioimmunoassay. Differences in all dependent variables between the trials will be determined using a repeated measures ANOVA and followed post-hoc when appropriate using paired T-tests to take advantage of the higher statistical power provided by paired comparisons. Data will be reported as means +/- SD. Significance will be selected at an alpha level of P < 0.05. These data may be useful as finding a snack source that produces a lower glycemic response and a greater satiating effect could be valuable in dietary counseling for blood glucose maintenance. For the cognitive portion of this research, these data may be useful because there is considerable room for improvement and for expanding evidence-based knowledge on the link between nutrition and cognition.

DETAILED DESCRIPTION:
Before each trial, subjects will fast for 10 hours. The 10-hour period of fasting is enough for development of the satiety index methodology. Subjects will be asked to refrain from caffeine and alcohol consumption, as well as strenuous exercise for the 32 hours prior to each blood collection. For both trials, participants will report to the lab at the same time each morning following the overnight fast. The subjects will report to the lab twice at least a week apart; once for the dried apple (240 kcal) trial and once the muffin (240 kcal) trial. After arriving at the lab, the participants will complete a cognitive pre-test (Concussion Vital Signs Test Battery) consisting of eight short cognitive tests on a computer. The cognitive pre- and post-tests will evaluate the following; verbal memory, visual memory, psychomotor speed, executive function, cognitive flexibility and reaction time. The participants will use their dominant hand to take the computerized test (except when indicated during the testing to use a specific hand during the "Finger Tapping Test") and will be asked to place their hand at the center of the space bar and keep their hand there during the cognitive testing. Participant's compliance and behaviors will be observed and noted by a research assistant. Next blood samples will be collected from warmed hands by finger-prick into large (250 microliter) heparinized Natelson tubes to obtain an ample blood collection for analysis of baseline plasma concentrations of glucose and insulin. Following baseline blood collection, subjects will rank their level of satiety and then consume the dried apple in their first visit to the lab and the muffin in their second visit to the lab. Subsequent blood samples and satiety ratings will be collected 15, 30, 45, 60, 90 and 120 minutes following the beginning of food consumption. Wash-out periods of at least a week between trials will allow for unbiased satiety index reporting by subjects. The satiety index of dried apple and muffin will be determined. Subjects will rate satiety on a 100 mm 7-point visual scale. Subjects will rank their level of satiety at any point along the scale. Participants will complete rankings on the scale prior to test food consumption and every 15 minutes after test food consumption. Participants will not have access to previously marked scales throughout the testing period. The developers of the satiety index have demonstrated that this scale provides greater retest reproducibility than a simple visual analog scale. Immediately after test food consumption, time required for food consumption will be recorded. Participants will answer the following questions using 100 mm visual analog scales (scale anchors indicated in parentheses). 1. How much did you like the meal? (0=Dislike extremely, 100=Like extremely) 2. How difficult was the food to eat? (0=Not at all difficult, 100=Extremely difficult) 3. Was the serving size sufficient? (0=Not at all enough, 100=Far too much) 4. How much more of this food would you like to eat? (0=Nothing at all, 100 A large amount) 5. Do you feel like eating something else? (0=Nothing at all, 100=A whole meal) 6. How much more food would you need to eat to completely satisfy your hunger? (0=Nothing at all, 100=A large amount) 7. Do you feel like eating something sweet (0=Not at all sweet, 100=Very sweet) 8. Do you feel like eating something salty (0=Not at all salty, 100=Very salty) 9. Do you feel like eating something savory (0=Not at all savory, 100=Very savory). Subjects will listen to a standardized playlist of music in between tests. Finally after the blood samples a satiety ratings are completed the participants will have a 10 minute break and then complete the cognitive post-test (Concussion Vital Signs Test Battery). The post-test will be a different version of the pre-test but the eight tests will remain in the same order for consistency. Prior to initiation of the study, an ample supply of dried apple and muffin will be obtained for the entire study. Collected blood will be centrifuged at 4°C to obtain plasma. Plasma will be stored in cryogenic vials at -70°C for batch analysis. Plasma glucose and insulin will be assessed at each time point. Glucose will be analyzed colorimetrically with kits from Stanbio Laboratory (Boerne, TX). Insulin will be determined using a radioimmunoassay from Diagnostics Products Corporation (Los Angeles, CA). The area under the glycemic response curve for the dried apple and muffin will be expressed relative to the mean response to glucose. Results will be reported as mean ± standard error of mean. Satiety index will be calculated as previously described as a measure of area under the curve for dried apple relative to muffin. Statistical analyses will be conducted using the Statistics Program for Social Sciences (SPSS) computer software package. Differences in glycemic index, satiety index, answers to visual analog scales, cognitive test scores and areas under the curve for biochemical parameters between different food trials will be determined using paired T-tests. Differences in other variables will be assessed with repeated measures ANOVAs and post-hoc paired T-tests as appropriate to take advantage of the higher statistical power provided by paired comparisons. Significance will be selected at an alpha level of P<0.05.

ELIGIBILITY:
Inclusion Criteria:

* Age: 20-45 years
* body mass index (BMI; in kg/m2): 18-25.

Exclusion Criteria:

* past head injuries,
* cigarette smoking,
* pregnancy,
* allergies to test foods,
* chronic use of medications known to affect metabolism,
* presence of any disorder or medications affecting metabolism (e.g., diabetes, hyperthyroidism, phenylketonuria, obesity, glycogen storage diseases, etc.).

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2015-09-23 (Actual); Primary Completion 2015-11-06 (Actual); Study Completion 2016-01-29 (Actual)

PRIMARY OUTCOMES:
blood glucose response | Changes from 0 to 120 minutes after consumption of test food
  blood glucose using reagent
serum insulin response | Changes from 0 to 120 minutes after consumption of test food
  serum insulin using ELISA

SECONDARY OUTCOMES:
various cognitive domains | baseline and two hour after test food consumption
  concussion vital signs test battery
Satiety | Changes from 0 to 120 minutes after consumption of test food
  Satiety using 100 mm 7 point visual scale

CONTACTS AND LOCATIONS:
Locations (1):
- San Diego State Univeristy, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No